CLINICAL TRIAL: NCT06905795
Title: Construction and Application of Full-cycle Screening and Mangement Techniques for MASLD in Children and Adolescents
Brief Title: Screening and Intervention of MASLD in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024S023
Record Dates: First submitted 2025-02-27; First posted 2025-04-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Children
Keywords: Children; MASLD; Lifestyle intervention; Screening

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comprehensive Intervention group (Experimental): Students in the comprehensive intervention group will receive the interventions including regular screening, nutrition guidance and increase physical activity lasting one year.
  Interventions: Diagnostic Test: Fibroscan test; Behavioral: Nutrition guidance; Behavioral: Increase physical activity; Other: Health education
- Monitoring Intervention group (Active Comparator): Students in the monitoring intervention group will receive regular sceeing every six months.
  Interventions: Diagnostic Test: Fibroscan test
- Control group (No Intervention): No Intervention.

INTERVENTIONS:
Diagnostic Test: Fibroscan test — Perform Fibroscan testing on the study subjects every six months.
  Arms: Comprehensive Intervention group; Monitoring Intervention group
Behavioral: Nutrition guidance — Each family will be matched with a nutritionist, who will provide daily online dietary guidance for parents and students during the first 21 days, followed by weekly sessions thereafter.
  Arms: Comprehensive Intervention group
Behavioral: Increase physical activity — Increase physical activity time in and out of school by professional sports trainer.
  Arms: Comprehensive Intervention group
Other: Health education — Knowledge of healthy lifestyle will be delivered in various forms such as health lectures, brochures, posters, etc.
  Arms: Comprehensive Intervention group

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) in children and adolescents has recently been renamed metabolic dysfunction-associated steatotic liver disease (MASLD). It has become one of the leading chronic liver diseases in children. The prevalence of MASLD is 6.3% among the general pediatric population and 40.4% among overweight and obese children, with an increasing trend each year. MASLD increases the risk of various metabolic diseases and can eventually lead to liver fibrosis or hepatocellular carcinoma, contributing to the disease burden.

Previous work by our project team using machine learning methods has identified that fasting insulin, alanine aminotransferase (ALT), and waist-to-height ratio (WHtR) have good predictive value in overweight and obese children, with a recommendation that children with a WHtR ≥ 0.48 should undergo further screening. However, external validation is still required to improve the effectiveness and cost-efficiency of this screening approach.

Till now, there are no approved drug treatments for paediatric MASLD, and lifestyle interventions (such as restricting energy intake and increasing physical activity) are the main therapeutic strategies. However, existing studies face limitations, such as small sample sizes, diverse intervention methods, lack of standardization, and short intervention durations, which hinder their clinical application. Therefore, it is essential to explore effective health lifestyle intervention models tailored to children.

This study aims to: First, optimizing the screening and treatment pathway, assess the cost-effectiveness and applicability of WHtR as a screening tool, and develop a tiered screening system suitable for Chinese children; Second, integrating school, clinic, family, and community resources to establish a multifacted lifestyle intervention model and evaluate its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* parents agree and support their children's weight loss, and students and parents have informed consent;
* students in two to four grade aged 7 and 11 years old;
* students with WHtR ≥ 0.48.

Exclusion Criteria:

* medical history of heart disease, hypertension, diabetes, tuberculosis, asthma, virus hepatitis or nephritis;
* obesity caused by endocrine diseases or side effects of drugs;
* abnormal physical development like dwarfism or gigantism;
* physical deformity such as severe scoliosis, pectus carinatum, limp, obvious O-leg or X-leg;
* inability to participate in school sport activities;
* a loss in weight by vomiting or taking drugs during the past 3 months.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Waist-to-Height Ratio | From enrollment to the end of treatment at 12 months and follow-up at 24 months

SECONDARY OUTCOMES:
Change in Controlled Attenuation Parameters | From enrollment to the end of treatment at 12 months and follow-up at 24 months
  Controlled Attenuation Parameters will be detected by Fibroscan HANDY
Change in Liver Stiffness Measurement | From enrollment to the end of treatment at 12 months and follow-up at 24 months
  Liver Stiffness Measurement will be detected by Fibroscan HANDY
Change in Blood Lipids | From enrollment to the end of treatment at 12 months
  Include TC, TG, LDL-C, and HDL-C
Change in Fasting Blood-Glucose | From enrollment to the end of treatment at 12 months
Change in Fasting Insulin | From enrollment to the end of treatment at 12 months
Change in Liver Enzyme | From enrollment to the end of treatment at 12 months
  Inlude ALT, AST, and GGT
Change in BMI | From enrollment to the end of treatment at 12 months and follow-up at 24 months
Change in BMI Z score | From enrollment to the end of treatment at 12 months and follow-up at 24 months
Change in Cardiorespiratory Endurance | From enrollment to the end of treatment at 12 months and follow-up at 24 months
  Cardiorespiratory Endurance will be assessed by 20 meter shuttle run test

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China